CLINICAL TRIAL: NCT04794829
Title: Natural History of Systemic and Nasal Mucosal Immunity to Influenza and SARS-CoV-2 in Adults After Vaccination
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000256; 000256-I
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09-10

CONDITIONS: Influenza; COVID-19
Keywords: Flu; Antibody; Immunization; Pandemic; COVID-19; Natural History
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinated: Received influenza and/or SARS-CoV-2 vaccine

SUMMARY:
Background:

Influenza (flu) vaccinations are required for all NIH staff members who have direct contact with patients. COVID-19 vaccines are recommended for persons 6 months of age and older. Researchers want to learn about immunity in NIH staff members who get a flu and/or COVID-19 vaccine.

Objective:

To understand what happens to the body s immune system throughout the year after getting the flu and/or COVID-19 vaccine.

Eligibility:

Adults ages 18 and older who work at NIH and plan to get the current season s flu vaccine and/or COVID-19 vaccine.

Design:

Participants will not get any vaccines as part of this study.

Participants will be screened with a medical history and medicine review. They will get a survey via email. It will ask about their flu and SARS-CoV-2 history and vaccinations.

Participants will have 12 monthly visits at NIH. If during that year they get both flu and SARS-COV-2 vaccines, their participation will be extended.

Once a month, participants will be contacted. They will discuss any new medicines, recent vaccinations, or changes in medical history.

Once a month, participants will have blood drawn.

Once a month, participants will have nasal sampling. A small, flat absorptive strip will be placed in the nostril to soak up mucus. Participants will press against the outside of their nostril with their finger for 1 minute.

Participants may be able to collect samples at home and mail them to NIH if they are not able to visit in person.

Participation will last for about 12 13 months.

DETAILED DESCRIPTION:
Study Description:

Yearly influenza vaccination is necessary due to short-lasting influenza immunity and changing strains of circulating influenza. With limited effectiveness of yearly influenza vaccines and the ongoing potential for an influenza pandemic, there is a need for a better understanding of influenza immunity to develop improved vaccines. Severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) vaccines have been developed in response to the coronavirus disease 2019 (COVID-19) pandemic. There is a critical need to also understand the changes in long-term immunity in those who receive a SARS CoV-2 vaccine to develop improved vaccines. We will investigate the changes in long-term immunity of NIH workers after vaccination with influenza and/or SARS-CoV-2 and throughout the following year via blood and nasal sampling.

Objectives:

Primary Objectives:

Characterize the systemic anti-influenza humoral immune response to vaccination over 1 year.

Characterize the systemic anti-SARS-CoV-2 humoral immune response to vaccination over 1 year.

Secondary Objectives:

Characterize the nasal mucosal anti-influenza humoral immune response to vaccination over 1 year.

Characterize the nasal mucosal anti-SARS-CoV-2 humoral immune response to vaccination over 1 year.

Endpoints:

Primary Endpoints:

1. Systemic anti-influenza antibodies as measured by:

   1. Hemagglutination inhibition (HAI) antibody titers
   2. Neuraminidase inhibition (NAI) antibody titers
   3. Anti-Hemagglutinin (HA) head antibody quantitative enzyme linked immunosorbent assay (ELISA) (immunoglobulin [Ig] M, IgG, IgA)
   4. Anti-HA stalk antibody quantitative ELISA (IgM, IgG, IgA)
   5. Anti-Neuraminidase (NA) antibody quantitative ELISA (IgM, IgG, IgA)
2. Systemic anti-SARS-CoV-2 antibodies as measured by:

   1. Anti-SARS-CoV-2 spike antibody quantitative ELISA (IgM, IgG, IgA)
   2. Anti-SARS-CoV-2 receptor binding domain (RBD) antibody quantitative ELISA (IgM, IgG, IgA)

Secondary Endpoints:

1. Mucosal anti-influenza antibodies from nasal samples as measured by:

   1. Anti-HA head antibody quantitative ELISA (IgA, IgG)
   2. Anti-HA stalk antibody quantitative ELISA (IgA, IgG)
   3. Anti-NA antibody quantitative ELISA (IgA, IgG)
2. Mucosal anti-SARS-CoV-2 antibodies from nasal samples as measured by:

   1. Anti-SARS-CoV-2 spike antibody quantitative ELISA (IgA, IgG)
   2. Anti-SARS-CoV-2 RBD antibody quantitative ELISA (IgA, IgG)

Study Population:

NIH staff (N=100) who are 18 years and older. NIH staff may include employees and contractors, fellows and volunteers. Accrual ceiling N=150.

Description of Sites/Facilities Enrolling Participants:

Participants will be enrolled at the NIH Clinical Center (CC).

Study Duration:

5 years

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. NIH staff members, at the time of enrollment.
2. Able to provide informed consent.
3. >=18 years of age.
4. Planning to receive the current influenza season s vaccine and/or an FDA-authorized or approved SARS-CoV-2 vaccine.
5. Willing and able to undergo blood draws or home blood samplings and nasal sampling procedures.
6. Willing and able to undergo at least one blood draw and one nasal sampling prior to receiving vaccine.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Already received the current season s influenza vaccine and does not plan to receive an FDA-authorized or approved SARS CoV-2 vaccine.
2. Already received an FDA-authorized or approved SARS-CoV-2 vaccine and does not plan to receive the current season s influenza vaccine.
3. Not willing to receive the current influenza season's vaccine and not willing to receive an FDA-authorized or approved SARS-CoV-2 vaccine.
4. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Co-enrollment guidelines: Participants may be co-enrolled in other studies; however, study staff should be notified of co-enrollment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NIH staff may include employees and contractors, fellows, and volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic anti-SARS-CoV-2 antibodies | One year
  Characterize the systemic anti SARS-CoV-2 humoral immune response to vaccination over 1 year.
Systemic anti-influenza antibodies | One year
  Characterize the systemic anti-influenza humoral immune response to vaccination over 1 year.

SECONDARY OUTCOMES:
Mucosal anti-SARS-CoV-2 antibodies from nasal samples | One year
  Characterize the nasal mucosal anti SARS-CoV-2 humoral immune response to vaccination over 1 year.
Mucosal anti-influenza antibodies from nasal samples | One year
  Characterize the nasal mucosal anti-influenza humoral immune response to vaccination over 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Han, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a small observational study, not an interventional trial. We will share data as currently outlined in the protocol.

REFERENCES:
- [Background] Black CL, Yue X, Ball SW, Fink RV, de Perio MA, Laney AS, Williams WW, Graitcer SB, Fiebelkorn AP, Lu PJ, Devlin R. Influenza Vaccination Coverage Among Health Care Personnel - United States, 2017-18 Influenza Season. MMWR Morb Mortal Wkly Rep. 2018 Sep 28;67(38):1050-1054. doi: 10.15585/mmwr.mm6738a2. PMID 30260944
- [Background] Ferdinands JM, Fry AM, Reynolds S, Petrie J, Flannery B, Jackson ML, Belongia EA. Intraseason waning of influenza vaccine protection: Evidence from the US Influenza Vaccine Effectiveness Network, 2011-12 through 2014-15. Clin Infect Dis. 2017 Mar 1;64(5):544-550. doi: 10.1093/cid/ciw816. Epub 2016 Dec 29. PMID 28039340
- [Background] Treanor JJ, Talbot HK, Ohmit SE, Coleman LA, Thompson MG, Cheng PY, Petrie JG, Lofthus G, Meece JK, Williams JV, Berman L, Breese Hall C, Monto AS, Griffin MR, Belongia E, Shay DK; US Flu-VE Network. Effectiveness of seasonal influenza vaccines in the United States during a season with circulation of all three vaccine strains. Clin Infect Dis. 2012 Oct;55(7):951-9. doi: 10.1093/cid/cis574. Epub 2012 Jul 25. PMID 22843783
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000256-I.html